CLINICAL TRIAL: NCT02508311
Title: The Effect of an Oral Beta-2 Agonist on Respiratory Muscle Strength in SCI
Brief Title: Albuterol to Improve Respiratory Strength in SCI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Our ability to test subjects with tetraplegia in this interventional study was interrupted by the COVID-19 pandemic. Our research pharmacist also informed us that oral albuterol is no longer being manufactured.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1910-P; SCH-15-011 (Other: James J. Peters Veterans Affairs Medical Center)
Record Dates: First submitted 2015-07-15; First posted 2015-07-24 (Estimated); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injury; Respiratory Muscle Weakness
Keywords: Tetraplegia; High Paraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Oral Beta-2 (Active Comparator): Subjects will receive 16 weeks of active medication.
  Interventions: Drug: Oral Albuterol Extended Release
- Placebo (Placebo Comparator): Subjects will receive 16 weeks of placebo medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Albuterol Extended Release — Subjects will receive extended release Albuterol, 4mg twice daily for the first week. The remaining 15 weeks subjects will receive extended release Albuterol, 8mg twice daily.
  Other Names: VoSpire
  Arms: Active Oral Beta-2
Drug: Placebo — Subjects will receive placebo tablets twice daily for 16 weeks.
  Arms: Placebo

SUMMARY:
Spinal cord injury (SCI), especially involving the cervical and upper thoracic segments, can significantly compromise respiratory muscle function. Respiratory complications can ensue, including lung collapse and pneumonia, which are the primary cause for mortality in association with traumatic SCI both during the acute and chronic phases post-injury. Lesions at the level of the cervical or high thoracic spinal cord result in respiratory muscle weakness, which is associated with ineffective cough, mucus retention, and mucus plugging. Despite the fact that pulmonary complications are a major cause of morbidity and mortality in this population, there is a paucity of effective interventions in the SCI population known to improve respiratory muscle strength with pharmacologic interventions receiving little to no attention. The current objective of this study is to determine the effectiveness of 16 weeks of sustained release oral Albuterol to; (1) improve respiratory muscular strength, and (2) improve cough effectiveness.

DETAILED DESCRIPTION:
Although the past 40 years has witnessed a substantial improvement in the acute and chronic management of persons with SCI, mortality remains high during the first year post-injury, and pulmonary complications including pneumonia, lung collapse (atelectasis), respiratory failure, and thromboembolism are the predominant cause. The propensity for pulmonary complications among subjects with SCI stems from paralysis of respiratory muscles. Injury to the cervical and upper thoracic cord significantly compromises function of the diaphragm, intercostal muscles, accessory respiratory muscles, and abdominal muscles. Respiratory muscle dysfunction is manifest as diminution in lung volumes, reduction in maximal static inspiratory and expiratory mouth pressures (MIP and MEP, respectively), and reduction in peak cough pressure and flow. Cough effectiveness is contingent upon both inspiratory and expiratory muscle strength; increasing the pressure-generating capacity of the inspiratory and expiratory muscles in persons with tetraplegia and high paraplegia may, therefore, translate to improved cough effectiveness and reduction in the propensity for atelectasis and, possibly, pneumonia.

Respiratory muscle training, often utilizing simple hand-held portable resistive or threshold training devices, appears to have marginal effects on vital capacity and maximal static mouth inspiratory and expiratory pressures (MIP and MEP, respectively), although data is inconclusive. Pharmacologic interventions to improve respiratory muscle strength have received little attention in the SCI population. Studies involving oral beta-2 adrenergic agonists, which have been shown to elicit anabolic effects on skeletal muscle in young men and an increase in muscle strength among patients with facioscapulohumeral muscular dystrophy, have also demonstrated salutary effects in persons with SCI. There are many foreseeable advantages of a pharmacologic approach to improve respiratory muscle strength in persons with SCI. For instance, RMT can be physically demanding and time consuming, compliance can be an issue, and sustainable improvements have not been realized. The intent in the present proposal is to enroll a targeted cohort of 24 comparatively weaker subjects with tetraplegia and high paraplegia in a randomized, double-blind, placebo-controlled, parallel group trial to assess the effects of an oral beta-2 agonist upon respiratory muscle strength and cough effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18 to 80
* Chronic spinal cord injury ( 1 year since injury)
* Neurological level of injury between C3-C8 (Tetraplegia)
* Neurological level of injury between T1-T6 (High Paraplegia)
* Males with maximal inspiratory pressure (MIP) < 90 cm H2O or
* Females with maximal inspiratory pressure (MIP) < 65 cm H2O

Exclusion Criteria:

* Smoking, active or history of smoking with the past year
* Ventilator Dependence
* History of blast injuries to the chest
* Antidepressant use
* History of asthma
* Active respiratory disease or recent(within 3 months) respiratory infections
* Uncontrolled hypertension or cardiovascular disease
* Current use a beta-2 adrenergic agonists
* History of epilepsy or seizure disorder
* Hyperthyroidism
* Currently taking corticosteroids
* Currently taking monoamine oxidase inhibitors or tricyclic antidepressants
* Hypersensitivity to albuterol or any of its' constituents
* Pregnant
* Use or are suspected of using over-the counter supplements or prescribed medications with anabolic characteristics (promotes improvements to muscle mass and strength) including, but not limited to:

  * creatine monohydrate
  * anabolic steroids (e.g., testosterone)
  * growth hormone
  * substances with similar actions or indications as those listed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Schilero, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD data is not available at this time.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Several participants failed screening, and thus were not randomized to either the treatment or placebo arm.
Period: Overall Study
Arm/Group | Active Oral Beta-2 | Placebo
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 9 participants screened, 1 participant was eligible; however, the participant withdrew. No data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Oral Beta-2 | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Respiratory Muscle Strength
Description: Respiratory muscle strength will be determined by maximal inspiratory pressure and maximal expiratory pressure at the mouth during baseline visit, week 16 visit and week 18 visit.
Time Frame: Baseline, Week 16, Week 18
Population: 1 participant screened and qualifies; however the participant dropped out. No data on this participant was collected.
Arm/Group | Active Oral Beta-2 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The one individual who consented and passed screening withdrew from the study prior to any data gathering, therefore no adverse events were reported.
Arm/Group | Active Oral Beta-2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Inability to perform study during COVID-19. Albuterol repetabs are also no longer being manufactured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT02508311/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT02508311/ICF_001.pdf